CLINICAL TRIAL: NCT07227077
Title: An Adaptive Design for Dosing Physical Activity Among Older Cancer Survivors Who Experience Chronic Pain: a Micro-randomized Trial
Brief Title: Dosing Physical Activity Among Older Cancer Survivors Who Experience Chronic Pain: a Micro-randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Whitney Morelli, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00055140; K01CA255414 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Cervical Cancer; Bladder Cancer; Colorectal Cancer; Endometrial Cancer; Lung Cancer; Prostate Cancer
Keywords: Physical Activity; Exercise; Survivorship; Supportive Care; Pain; Symptom Management
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Micro-Randomized Trial (MRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micro-randomized trial study arm (Experimental): In this one-armed, 4-week trial, participants will receive prompts to report their pain symptoms 4 times throughout the day. Participants may receive up to 4 reminders to move messages throughout the day to promote participants to engage in physical activity. The receipt of messages is randomized each day. Participants will wear a research-grade activity monitor throughout the duration of their participation in the intervention to measure physical activity behaviors.
  Interventions: Behavioral: Physical Activity Promotion Intervention

INTERVENTIONS:
Behavioral: Physical Activity Promotion Intervention — This physical activity promotion intervention is a micro-randomized trial designed to determine the most effective time to send a message to promote physical activity among cancer survivors who experience chronic pain symptoms.

SUMMARY:
The purpose of this study is to assess the best time to deliver a message to increase physical activity and how often participants will experience a pain episode in the 24 hours following their receipt of a message to increase physical activity.

DETAILED DESCRIPTION:
The primary objective of this study is to test a theory-based, micro-randomized trial to determine the optimal state to deliver a message to increase physical activity by determining the probability older cancer survivors will be physically active in the one hour following a messaging prompt. The secondary, exploratory objective is to determine the probability older cancer survivors will experience a pain episode in the 24 hours following their receipt of a message to increase physical activity.

Eligibility criteria is deliberately incomplete to preserve the scientific integrity of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 65 years.
2. Patients with a history of bladder, breast, cervical, colorectal, endometrial, lung, and prostate cancer diagnosis and treatment.
3. Fluent in spoken and written English.
4. Patient has access to smartphone
5. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Patient has metastatic disease.
2. Patient has cancer recurrence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
ActiGraph accelerometer measured physical activity behaviors (sedentary, light, moderate, vigorous intensity). | 4 weeks
  Physical activity will be measured using an ActiGraph accelerometer. Data will be aggregated into physical activity estimations (sedentary, light, moderate, vigorous, steps, etc.) using standard methods. Outcome of interest will be probability older cancer survivors are physically active in the 30 minutes following the receipt of a messaging prompt to promote physical activity.
11-point box scale to assess pain on a scale of 0 (no pain) to 10 (worst possible pain). | 4 weeks
  Pain state will be assessed by response to the pain rating measured by the 11-Point Box Scale in the study app. Participants will receive a smart phone prompt to rate their pain 4 times per day. Outcome of interest will be probability older cancer survivors experience a pain episode in the 24 hours following the receipt of a messaging prompt to increase physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No